CLINICAL TRIAL: NCT07053384
Title: An Exploratory Phase 1b, Multicenter, Randomized, Open-Label Study to Investigate the Impact of the Administration of Intravenous VH3810109 With or Without Oral Fostemsavir in Combination With Integrase Inhibitor-Based Antiretroviral Therapy on the Viral Reservoir in Adults Living With HIV-1
Brief Title: A Study to Investigate the Use of VH3810109 With or Without Fostemsavir (FTR) to Reduce the Size and Activity of the Viral Reservoir in People Living With HIV
Acronym: ENTRANCE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221794; 2025-520629-19-00 (Other: EU CT Number)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: VH3810109; N6LS; Broadly neutralizing antibody (bNAb); Fostemsavir (FTR); RUKOBIA; INSTI-based ART; Human Immunodeficiency Virus (HIV); HIV reservoir; Adults living with HIV
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants receiving standard of care (SOC) integrase strand transfer inhibitor (INSTI)-based ART (Active Comparator)
  Interventions: Drug: SOC INSTI-based ART
- Participants receiving SOC INSTI-based ART plus VH3810109 (Experimental)
  Interventions: Biological: VH3810109; Drug: SOC INSTI-based ART
- Participants receiving SOC INSTI-based ART plus VH3810109 plus FTR (Experimental)
  Interventions: Biological: VH3810109; Drug: Fostemsavir (FTR); Drug: SOC INSTI-based ART

INTERVENTIONS:
Biological: VH3810109 — VH3810109 will be administered.
  Arms: Participants receiving SOC INSTI-based ART plus VH3810109; Participants receiving SOC INSTI-based ART plus VH3810109 plus FTR
Drug: Fostemsavir (FTR) — Fostemsavir will be administered.
  Other Names: RUKOBIA
  Arms: Participants receiving SOC INSTI-based ART plus VH3810109 plus FTR
Drug: SOC INSTI-based ART — A SOC INSTI-based ART regimen will be administered.

SUMMARY:
This study investigates the use of VH3810109 with or without FTR to reduce the size and activity of the HIV viral reservoir in two sub-populations of people living with HIV: treatment-naïve adults (Population 1) and treatment-experienced adults currently taking a standard of care (SOC) integrase strand transfer inhibitor (INSTI)-based antiretroviral therapy (ART) regimen (Population 2).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 70 years old at the time of obtaining informed consent.
* Persons of any sex or gender are eligible. Note: Participants of childbearing potential (POCBP) are eligible to participate if not pregnant, not lactating, and agreeing to adhere to study requirements for use of contraception and pregnancy avoidance.
* Participant has a documented diagnosis of HIV-1 infection Note: Participants in Population 1 must have a documented positive HIV antibody result available for Screening.

Population 1 only:

* Plasma HIV-1 RNA >=2000 copies/milliliter (c/mL) at Screening.
* CD4+ T cell count >=300 cells/microliter (μL) at Screening.
* Antiretroviral treatment naïve, defined as no exposure to ART after a diagnosis of HIV-1 infection, prior to enrollment.

Population 2 only:

* Participant is stably virologically suppressed (plasma HIV-1 RNA <50 c/mL).
* Documented evidence of uninterrupted treatment with oral non-boosted INSTI-based ART for at least 6 months prior to Screening, as well as uninterrupted treatment with ART (any guideline-recommended oral regimen) for at least 24 months prior to Screening.
* CD4+ T cell count >=450 cells/μL at Screening.
* Body weight >=50 kg to <=115 kg.
* Participant is capable of giving written informed consent, which includes adherence to the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

CONCURRENT MEDICAL CONDITIONS & MEDICAL HISTORY

* Participant is pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.
* Participant has documented diagnosis of HIV-2 infection.
* Participant is known to have acquired HIV via perinatal transmission.
* Any evidence of a current or known past Center for Disease Control and Prevention (CDC) Stage 3 disease.
* Any ongoing malignancy or history of systemic cancers, such as Kaposi's sarcoma and lymphoma, or other virus-associated malignancies.
* Ongoing or clinically relevant pancreatitis.
* Current HIV-related kidney disease.
* History of or active HIV-associated dementia or progressive multifocal leukoencephalopathy.

CARDIAC & CARDIOVASCULAR CONDITIONS

• Participants who are at clinically significant risk of cardiovascular disease.

* Ongoing or any lifetime history of clinically significant cardiovascular or cardiac disease.
* Confirmed QTcF value outside normal range at Screening or Day 1.

HEPATIC CONDITIONS

• History of clinically relevant hepatitis in the 6 months prior to Screening.

* Participants with severe hepatic impairment.
* Advanced MAFLD and advanced non-alcoholic steatohepatitis, if evidence for substantial fibrosis (fibrosis score ≥F2) or evidence of cirrhosis.
* Unstable liver disease.
* History of liver cirrhosis with or without hepatitis viral co-infection.

NEUROPSYCHIATRIC CONDITIONS

• Participants who pose a significant suicide risk.

LABORATORY DIAGNOSTIC ASSESSMENTS

* Participants who are experiencing (Population 1) or are known to have initiated ART during (Population 2) acute HIV infection.
* Any verified Grade 4 laboratory abnormality at Screening, excluding asymptomatic elevations of lipids or CPK.
* Alanine transferase (ALT) >=3 times the upper limit of normal (ULN) at Screening.
* Estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73 m^2.
* Hemoglobin >=Grade 2 at Screening.
* Platelets >=Grade 2 at Screening.
* Absolute Neutrophil Count (ANC) ≥Grade 2 at Screening.
* Any acute abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's inclusion in an interventional clinical study.

Population 2 only • Two or more plasma HIV-1 RNA results >=50 c/mL in the 18 months prior to Screening.

INFECTIOUS DISEASES

* Active hepatitis B virus (HBV) co-infection.
* Active hepatitis C virus (HCV) co-infection.
* Participant has untreated syphilis before enrolment.
* Known current untreated or incompletely treated active Mycobacterium TB infection.

ANTIRETROVIRAL RESISTANCE

• Known major resistance-associated mutations to second-generation INSTIs or to antiretroviral (ARV) agents from 2 or more drug classes.

PRIOR AND CONCOMITANT MEDICATIONS

* Prior use of any of the following agents:

  o long-acting ARVs (any dose in the past 24 months or within 5 half-lives [whichever is longer])

  o FTR (any lifetime use)
  * HIV-1 immunotherapeutic vaccines or prophylactic vaccines (any lifetime use)
  * HIV-1 monoclonal antibody therapy (any lifetime use).
* Prior receipt of any approved or experimental non-HIV vaccination within 2 weeks prior to study enrolment.
* History of systemic corticosteroids, immunosuppressive anti-cancer, interleukins, systemic interferons, or systemic chemotherapy, within 6 months prior to Screening.
* Participant has received an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent (whichever is longer), prior to enrolment.
* Treatment with any of the following agents within 30 days of enrolment:

  o radiation therapy

  o cytotoxic chemotherapeutic agents
  * anti-tuberculosis therapy
  * immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons.
* Participant is receiving any protocol-defined prohibited medication and is unwilling or unable to switch to an alternate medication. Prohibited medications must be stopped within 7 days (or 14 days if the drug is a potential CYP3A4 enzyme inducer) or 5 half-lives (whichever is longer), prior to enrolment.

Population 1 only • Known use of PrEP or PEP within <30 days (for oral agents) or <52 weeks (for LA parenteral agents) of HIV-1 diagnosis. Participants with a documented seronegative result >=30 days after the last dose of oral PrEP or PEP (or >=52 weeks after the last dose of LA PrEP) are not excluded.

Population 2 only

• Current use of NNRTI-containing ART.

OTHER EXCLUSIONS

* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class, or a history of drug or other allergy that contraindicates study participation.
* Any condition which may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study drugs.
* Any pre-existing physical or mental condition (including substance use disorder) which, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participant is currently participating in, or anticipates being selected for, any other interventional study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2028-03-24 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cell-associated HIV-1 RNA transcripts per million cluster of differentiation 4 (CD4+) T cells | From Baseline (Day 1) to Month 12

SECONDARY OUTCOMES:
Change from baseline in total, intact, and defective proviral HIV-1 DNA per million CD4+ T cells | From Baseline (Day 1) to Month 12
Absolute change in cell-associated HIV-1 RNA/proviral DNA ratios in CD4+ T cells | From Baseline (Day 1) to Month 12
Absolute values for p24+ CD4+ T cell count | From Baseline (Day 1) to Month 12
Change from baseline in number of p24+ CD4+ T cells | From Baseline (Day 1) to Month 12
Absolute values for HIV-1-specific CD8+ T cell count | From Baseline (Day 1) to Month 12
Change from baseline in HIV-1-specific CD8+ T cell count | From Baseline (Day 1) to Month 12
Number of participants with Grade 3 and Grade 4 adverse events (AEs) | From Baseline (Day 1) to Month 12
Number of participants with serious adverse events (SAEs), deaths and AEs leading to discontinuation of study intervention | From Baseline (Day 1) to Month 12

CONTACTS AND LOCATIONS:
Locations (25):
- United States (12):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- Denmark (2):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Hvidovre
- GSK Investigational Site, Rotterdam, Netherlands
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, La Laguna Santa Cruz
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf